CLINICAL TRIAL: NCT02668380
Title: An Open Label, Prospective, Multicentre, Non-interventional Study of Apatinib for Chemotherapy-Refractory Advanced Metastatic Gastric Cancer
Acronym: AHEAD-G202
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AHEAD-G202
Record Dates: First submitted 2015-12-05; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Gastric Cancer
Keywords: Apatinib; metastatic gastric cancer; Non-interventionalStudy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Apatinib: Apatinib Tablets: 850 mg,po, once daily , 28 days for a cycle

SUMMARY:
This is an Open Label, Prospective, Multicentre, Non-interventional Study of Apatinib for Chemotherapy-Refractory Advanced Metastatic Gastric Cancer, the investigators opted to give patients for apatinib 850 mg once daily, 28 days for a cycle. To evaluate the safety and efficacy of apatinib for Advanced Metastatic Gastric Cancer in the real world.

DETAILED DESCRIPTION:
In the last decade, front-line chemotherapy has been considered a standard therapeutic regimen for the extension of survival time in patients with metastatic gastric cancer (mGC). New evidence suggests that salvage chemo-therapies, as second-line treatments, may have a survival advantage when compared with best supportive care. After failure of second-line chemotherapy, the results of further treatment are poor, yielding response rates of 0% to 5% with no evidence of prolonged survival. Apatinib is a small-molecule VEGFR-2 tyrosine kinase inhibitor, Had been approved by the CFDA for the treatment of advanced gastric cancer, However, this study defines a variety of inclusion/exclusion criteria, efficacy and safety are not well reflect in the real world for the treatment of advanced gastric cancer. Therefore, an Open Label, Prospective, Multicentre, Non-interventional Study could evaluate the safety and efficacy of apatinib for Advanced Metastatic Gastric Cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

* 》18 years old
* Advanced Metastatic Gastric Cancer
* The doctor evaluate that patients had benefit from treatment
* The patients signed the written informed consent

Exclusion Criteria:

* Apatinib has been confirmed for allergy sufferers
* Pregnant or lactating women
* Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, within 30 days after major surgery, uncontrolled high blood pressure medication, III-IV level cardiac insufficiency, severe liver and kidney dysfunction)
* Doctors think doesn't inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Metastatic Gastric Cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 1 years
  Treatment-related toxicities were graded according to Common Terminology Criteria Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Overall survival | 1 years
  Overall survival (OS) was calculated from the date of initial treatment with apatinib to the date of death due to any cause.
Progression-free survival | 8 months
  A duration from the date of initial treatment with apatinib to disease progression(as defined by RECIST) or death.
Objective response rate | 5 months
  Number of participants who achieve complete response or partial response. Either complete response (CR) or partial response (PR) will be evaluated by RECIST, confirmed at least 4 weeks following the date of the initial response.

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Oncology and Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li N, Bai C, Zhang R, Ma L, Ren X, Zhang J, Fu Z, Zhao L. Efficacy and safety of apatinib for the treatment of AFP-producing gastric cancer. Transl Oncol. 2021 Feb;14(2):101004. doi: 10.1016/j.tranon.2020.101004. Epub 2020 Dec 28. PMID 33383486
- [Derived] Wang X, Zhang R, Du N, Yang M, Zang A, Liu L, Yu J, Gao J, Zhang J, Fu Z, Ren Y, Ma L, Guo J, Li Q, Li X, Fan Z, Song X, Liu Z, Zhang Y, Li G, Yu Z, Diao J, Jia J, Liang F, Wang H, Sun J, Gao Y, Yang P, Bai C, Ren X, Zhong D. An open label, multicenter, noninterventional study of apatinib in advanced gastric cancer patients (AHEAD-G202). Ther Adv Med Oncol. 2020 Mar 19;12:1758835920905424. doi: 10.1177/1758835920905424. eCollection 2020. PMID 32218807